CLINICAL TRIAL: NCT07345468
Title: Fear of Childbirth, Birth Beliefs, Mode of Birth Preferences in Pregnants' Participating in Childbirth Preparation Classes: A Quasi-Experimental Study
Brief Title: Fear of Childbirth, Birth Beliefs, Mode of Birth Preferences in Childbirth Preparation Classes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Sevil Cicek Ozdemir, Principal Investigator, Kutahya Health Sciences University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KutahyaHSUU
Record Dates: First submitted 2025-09-24; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Fear of Childbirth; Beliefs About Childbirth; Mode of Birth; Childbirth Preparation Classes
Keywords: Childbirth; Fear; Education; Nursing; Parturition; Pregnancy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- face-to-face childbirth preparation classes (Other): The training was given face-to-face in the face-to-face classes group
  Interventions: Other: face-to-face childbirth preparation education
- online childbirth preparation classes (Other): The training was given online in the online classes group.
  Interventions: Other: online childbirth preparation education

INTERVENTIONS:
Other: face-to-face childbirth preparation education — Women in the face-to-face education group received face-to-face childbirth preparation classes.
  Arms: face-to-face childbirth preparation classes
Other: online childbirth preparation education — Women in the online group received online classes at the same time.
  Arms: online childbirth preparation classes

SUMMARY:
Objective: The aim of this research study is to evaluate the fear of childbirth, birth beliefs, and mode of birth preferences in pregnant who participated in face-to-face and online childbirth preparation classes.

Method: This research is a quasi-experimental study. Pregnant will assign to two intervention groups, face-to-face, and online childbirth preparation classes. Data will collected twice, before (pre-test) and one-month after (post-test) the childbirth preparation training. The training will give face-to-face in the face-to-face classes group. The training will give online in the online classes group.

DETAILED DESCRIPTION:
Teaching techniques such as presentation, question and answer, games, group discussion, and animation videos are used in the sessions. In addition, exercises such as massage, breathing, and relaxation exercises are practiced together.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-45 years
* Nulliparous,
* First and singleton pregnancy,
* Between 20-32 weeks of gestation,
* Without any pregnancy-related risk factors,
* Who had not participated in any other childbirth preparation training,
* Had at least a primary education level, had no communication difficulties,
* Had access to and were able to use an internet-connected device with a camera.

Exclusion Criteria:

* Multiparous pregnant who had multiple pregnancies,
* Had any high-risk pregnancy symptoms,
* Were below the 20th week and above the 32nd week.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2023-07-15 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
fear of childbirth | before (pre-test) and one-month after (post-test) the childbirth preparation training
  Level of childbirth fear
birth beliefs | before (pre-test) and one-month after (post-test) the childbirth preparation training
  Natural or medical birth beliefs
mode of birth preferences | before (pre-test) and one-month after (post-test) the childbirth preparation training
  Preferred mode of birth

CONTACTS AND LOCATIONS:
Locations (1):
- Kütahya Health Sciences University, Kütahya, Turkey (Türkiye)